CLINICAL TRIAL: NCT07215182
Title: [68Ga]Ga-FAPI PET/CT for Response Evaluation During Immune Checkpoint Inhibitor Therapy in Malignant Melanoma
Brief Title: [68Ga]Ga-FAPI Total Body PET/CT for Better and Faster Imaging in Cancer
Acronym: BEFAST
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Barbara Malene Fischer (Other)
Collaborators: Herlev Hospital (Other)
Responsible Party: Sponsor-Investigator, Barbara Malene Fischer, Professor, MD, Ph.D., Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 522_22; 2023-509549-11-00 (EU CTIS Number)
Record Dates: First submitted 2025-09-10; First posted 2025-10-10 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Malignant Melanoma Stage IV
Keywords: FAPI PET/CT; Immune checkpoint inhibitor therapy; malignant melanoma; response evaluation
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Masking Description: The baseline and the follow-up [68Ga]Ga-FAPI-46 PET/CT scan will be evaluated by a team of experienced specialists in clinical physiology and nuclear medicine, and radiology. These specialists are blinded from findings on the standard imaging ([18F]FDG PET/CT).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Advanced staged Malignant Melanoma (Experimental): Patients with advanced stage malignant melanoma with visible lesions on [18F]FDG PET/CT referred for ICT at the Dept. of Oncology Herlev Hospital will be sought enrolled. Patients will undergo two [68Ga]Ga-FAPI-46 PET/CT, which include injection with the experimental tracer [68Ga]Ga-FAPI-46. These scans are in addition to their standard imaging.
  Interventions: Drug: [68Ga]Ga-FAPI-46

INTERVENTIONS:
Drug: [68Ga]Ga-FAPI-46 — Patients undergo two PET/CTs with the experimental tracer [68Ga]Ga-FAPI-46 (drug).

SUMMARY:
The goal of this clinical trial is to investigate the use of the tracer [68Ga]Ga-FAPI-46 for PET/CT-imaging in response evaluation of patients with advanced stage malignant melanoma treated with immune checkpoint inhibitor therapy (ICT). The main question it aims to answer is:

• Can [68Ga]Ga-FAPI-46 PET/CT improve response evaluation in patients suffering from advanced stage malignant melanoma treated with ICT and potentially serve as a biomarker.

Researchers will compare findings on the experimental [68Ga]Ga-FAPI-46 PET/CT with findings on standard imaging ([18F]FDG PET/CT).

Participants will undergo:

* Two [68Ga]Ga-FAPI-46 PET/CT scans: one before treatment initiation with ICT and one after three months.
* Two blood samples
* Passive follow-up 6 months after the last scan [68Ga]Ga-FAPI-46 PET/CT

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, >/=18 years old
2. Histological verified metastatic or locally advanced malignant melanoma
3. Visible malignant lesions on [18F]FDG PET/CT or CT
4. Subjects must be considered inoperable
5. Subjects must be considered medically suitable for ICT
6. Subjects must be able to read and understand the patient information in Danish to give informed consent

Exclusion Criteria:

1. Ocular or mucosal melanoma
2. Other concurrent cancer disease
3. Previous systemic oncological treatment with ICT
4. Pregnancy or lactation
5. Weight more than the maximum limit of a PET/CT-scanner bed (140 kg)
6. History of allergic reaction due to compounds similar to the chemical composition of [68Ga]Ga-FAPI- 46

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-08-15 (Actual); Primary Completion 2026-08-20 (Estimated); Study Completion 2027-02-20 (Estimated)

PRIMARY OUTCOMES:
Changes in FAPI-uptake in malignant lesions on [68Ga]Ga-FAPI-46 PET/CT during ICT | From enrollment in the study (signed informed consent) to after the second [68Ga]Ga- FAPI PET/CT, estimated time is 3 months.
  Specified malignant lesions will be defined and evaluated by a team of specialists on the baseline [68Ga]Ga- FAPI PET/CT scan and the uptake of the FAPI tracer in the lesions will be quantified. The evaluation of the malignant lesions on [68Ga]Ga-FAPI PET/CT will also be compared with a similar lesion evaluation on the [18F]FDG PET/CT (standard imaging). The FAPI-uptake will be reassessed after 12 weeks of ICT by the same team of specialists. Changes in uptake of malignant lesions after 12 weeks of ICT on the [68Ga]Ga-FAPI-46 PET/CT will be compared to changes on the [18F]FDG PET/CT and the clinical response. The clinical response will be assessed using the patients' medical record.

SECONDARY OUTCOMES:
Changes in [68Ga]Ga-FAPI-46-uptake during ICT in healthy tissue | From enrollment in the study (signed informed consent) to the end of the follow-up (6 months after the second [68Ga]Ga-FAPI-46 PET/CT, estimated time in total is 9 months from signed informed consent).
  Tracer-uptake in healthy tissue and benign lesions on [68Ga]Ga-FAPI-46 PET/CT will be evaluated using the same method as described in "Primary Objectives". A similar evaluation of standard [18F]FDG PET/CT will be performed. FAPI-uptake in healthy tissue on [68Ga]Ga-FAPI-46 PET/CT will be compared to the findings on [18F]FDG PET/CT. To verify the [68Ga]Ga-FAPI-46 PET/CT assessment (including evaluation of healthy tissue, malignant lesions and benign lesions), the assessment will be compared to the findings from a composed reference standard. This consist of all available imaging, biopsy results, blood tests, and information on hospitalization and changes in patient management up to 6 months after the [68Ga]Ga-FAPI PET/CT.

OTHER OUTCOMES:
Correlation between [68Ga]Ga-FAPI-46-uptake on [68Ga]Ga-FAPI-46 PET/CT and levels of FAP-activity biomarkers in serum blood samples during ICT. | From enrollment in the study (signed informed consent) to the end of the follow-up (6 months after the second [68Ga]Ga-FAPI-46 PET/CT, estimated time in total is 9 months from signed informed consent).
  Blood samples from the included participants will be analyzed by Nordic Bioscience- Results from this analysis will be correlated to the disease activity evaluated on the [68Ga]Ga-FAPI-46 PET/CT. Results from the serum blood sample analysis will also be correlated with treatment outcome after 6 months of treatment. Treatment outcome will be defined using the RECIST criteria (40). This analysis will be done retrospectively on routine clinical scans ([18F]FDGPET/CT). The updated guideline and definitions of the RECIST criteria will be used.

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Herlev Universityhospital, Herlev, Capital Region
  - Rigshospitalet, Copenhagen, Ca

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zhang HE, Hamson EJ, Koczorowska MM, Tholen S, Chowdhury S, Bailey CG, Lay AJ, Twigg SM, Lee Q, Roediger B, Biniossek ML, O'Rourke MB, McCaughan GW, Keane FM, Schilling O, Gorrell MD. Identification of Novel Natural Substrates of Fibroblast Activation Protein-alpha by Differential Degradomics and Proteomics. Mol Cell Proteomics. 2019 Jan;18(1):65-85. doi: 10.1074/mcp.RA118.001046. Epub 2018 Sep 26. PMID 30257879
- [Background] Ferdinandus J, Kessler L, Hirmas N, Trajkovic-Arsic M, Hamacher R, Umutlu L, Nader M, Zarrad F, Weber M, Fendler WP. Equivalent tumor detection for early and late FAPI-46 PET acquisition. Eur J Nucl Med Mol Imaging. 2021 Sep;48(10):3221-3227. doi: 10.1007/s00259-021-05266-7. Epub 2021 Feb 23. PMID 33620560
- [Background] Hirmas N, Hamacher R, Sraieb M, Ingenwerth M, Kessler L, Pabst KM, Barbato F, Lueckerath K, Kasper S, Nader M, Schildhaus HU, Kesch C, von Tresckow B, Hanoun C, Hautzel H, Aigner C, Glas M, Stuschke M, Kummel S, Harter P, Lugnier C, Uhl W, Niedergethmann M, Hadaschik B, Grunwald V, Siveke JT, Herrmann K, Fendler WP. Fibroblast-Activation Protein PET and Histopathology in a Single-Center Database of 324 Patients and 21 Tumor Entities. J Nucl Med. 2023 May;64(5):711-716. doi: 10.2967/jnumed.122.264689. Epub 2022 Dec 29. PMID 36581374
- [Background] Meyer C, Dahlbom M, Lindner T, Vauclin S, Mona C, Slavik R, Czernin J, Haberkorn U, Calais J. Radiation Dosimetry and Biodistribution of 68Ga-FAPI-46 PET Imaging in Cancer Patients. J Nucl Med. 2020 Aug;61(8):1171-1177. doi: 10.2967/jnumed.119.236786. Epub 2019 Dec 13. PMID 31836685
- [Background] Finke D, Heckmann MB, Herpel E, Katus HA, Haberkorn U, Leuschner F, Lehmann LH. Early Detection of Checkpoint Inhibitor-Associated Myocarditis Using 68Ga-FAPI PET/CT. Front Cardiovasc Med. 2021 Feb 25;8:614997. doi: 10.3389/fcvm.2021.614997. eCollection 2021. PMID 33718446
- [Background] Hotta M, Sonni I, Benz MR, Gafita A, Bahri S, Shuch BM, Yu R, Liu ST, Czernin J, Calais J. 68Ga-FAPI-46 and 18F-FDG PET/CT in a patient with immune-related thyroiditis induced by immune checkpoint inhibitors. Eur J Nucl Med Mol Imaging. 2021 Oct;48(11):3736-3737. doi: 10.1007/s00259-021-05373-5. Epub 2021 Apr 29. No abstract available. PMID 33914106
- [Background] Rong X, Lv J, Liu Y, Wang Z, Zeng D, Li Y, Li S, Wu J, Shen Z, Shi M, Liao W, Wu Z, Wang C. PET/CT Imaging of Activated Cancer-Associated Fibroblasts Predict Response to PD-1 Blockade in Gastric Cancer Patients. Front Oncol. 2022 Jan 26;11:802257. doi: 10.3389/fonc.2021.802257. eCollection 2021. PMID 35155199
- [Background] Monteran L, Erez N. The Dark Side of Fibroblasts: Cancer-Associated Fibroblasts as Mediators of Immunosuppression in the Tumor Microenvironment. Front Immunol. 2019 Aug 2;10:1835. doi: 10.3389/fimmu.2019.01835. eCollection 2019. PMID 31428105
- [Background] Mokoala K, Emil N, Lawal I, Antke C, Giesel FL, Sathekge M. [68 Ga]Ga-FAPI versus [18F]F-FDG in malignant melanoma: complementary or counterpoint? Eur J Nucl Med Mol Imaging. 2022 Jun;49(7):2445-2446. doi: 10.1007/s00259-022-05702-2. Epub 2022 Feb 9. No abstract available. PMID 35137262
- [Background] Zhou L, Yang K, Andl T, Wickett RR, Zhang Y. Perspective of Targeting Cancer-Associated Fibroblasts in Melanoma. J Cancer. 2015 Jun 23;6(8):717-26. doi: 10.7150/jca.10865. eCollection 2015. PMID 26185533
- [Background] Nurmik M, Ullmann P, Rodriguez F, Haan S, Letellier E. In search of definitions: Cancer-associated fibroblasts and their markers. Int J Cancer. 2020 Feb 15;146(4):895-905. doi: 10.1002/ijc.32193. Epub 2019 Feb 28. PMID 30734283

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-06-02): https://cdn.clinicaltrials.gov/large-docs/82/NCT07215182/Prot_SAP_000.pdf
  • Informed Consent Form (2025-02-01): https://cdn.clinicaltrials.gov/large-docs/82/NCT07215182/ICF_001.pdf